CLINICAL TRIAL: NCT00708318
Title: A Pilot, Phase I, 2-Period, Fasting, Bioavailability, Safety and PK Study Evaluating A Single Dose Intravenous Fentanyl 200 µg) and Single Doses of 2 or 3 mL AeroLEF (Liposome-Encapsulated Fentanyl 500 µg/mL) in Normal Healthy Non Subjects
Brief Title: Study Evaluating Inhaled AeroLEF (Liposome-Encapsulated Fentanyl)in Normal Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Responsible Party: Ali Raza, Chief Medical Officer, YM BioSciences
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEF-2494
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: AeroLEF; fentanyl; pharmacokinetic; liposome; encapsulated
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A, B, C (Experimental)
  Interventions: Drug: i.v. fentanyl and AeroLEF

INTERVENTIONS:
Drug: i.v. fentanyl and AeroLEF — Period I: subjects received an intravenous dose of fentanyl (200 µg) (Treatment A).
  Period II: subjects were randomly assigned to receive either 2 mL (Treatment B) or 3mL (Treatment C) of AeroLEF delivered by nebulization with an AeroEclipse BAN.
  Other Names: Ionsys; Depodur; fetanyl

SUMMARY:
This was a pilot, phase I, two-period, fasting, bioavailability, safety,and pharmacokinetic study evaluating single dose of i.v. fentanyl (200 µg) and single doses of 2 mL or 3 mL inhaled AeroLEF (500 µg/mL) delivered by nebulization with the AeroEclipse BAN device administered in normal healthy non-smoking subjects.

DETAILED DESCRIPTION:
In Period I, subjects received an intravenous dose of fentanyl (200 µg) administered over 1 minute (Treatment A). Subjects then crossed over to Period II.

In Period II, subjects were randomly assigned to receive either 2 mL (1000 µg fentanyl; Treatment B) or 3mL (1500 µg fentanyl; Treatment C) of AeroLEF delivered by nebulization with the AeroEclipse BAN. Subjects were instructed to continue inhalation of AeroLEF for approximately 1 minute beyond the point of nebulizer sputter to ensure that all aerosolized medication was delivered. There was at least a 1 week washout period between study periods.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female with a minimum age of at least 18 years
* Body weight with aBMI range of 18.5 - 27, with a minimum weight of at least 60 kg.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed, written, Informed Consent Form.
* Normal findings in the physical examination, vital signs (blood pressure between 100-140 - 60-90 mmHg, heart rate between 55-99 beats/min, respiration rate between 12-20 minute) and a 12 lead ECG.
* Negative for drug abuse, nicotine, alcohol, hepatitis B-surface antigen, hepatitis C and HIV.
* If a female of child-bearing potential, the patient must have a negative urine pregnancy test at screening and baseline.
* No clinical laboratory values outside of the Principal Investigator's acceptable range, unless the Principal Investigator decided that the subject's values are not clinically significant.
* Female subjects: (a) if pre-menopausal, have regular menstrual cycles (28-32 days), and (b) are not pregnant prior to study start and avoids pregnancy during the study and 1 month post drug administration, or (c) were surgically sterile for at least 6 months prior to enrollment, or (d) are post-menopausal for at least 1 year prior to enrollment.

Exclusion Criteria:

* Known history of hypersensitivity to fentanyl.
* Presence or history of cardiac, pulmonary, gastrointestinal, endocrine, neuromuscular, neurologic, hematological, liver or kidney disease, or any condition known to interfere with absorption, distribution , metabolism, or excretion of drugs.
* History of drug abuse or narcotic dependency.
* Use of prescription medication within 30 days preceding entry int the study, including any enzyme inducing/inhibitory drugs (excluding contraceptives).
* Participating in a clinical trial with an investigational drug within 30 days preceding this trial.
* Blood donation within 45 days preceding this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2001-10; Primary Completion 2001-11 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | continuously

SECONDARY OUTCOMES:
pharmacokinetics | various time points

CONTACTS AND LOCATIONS:
Overall Officials: Diana Pilura, PhD, Study Director — YM BioSciences; Paul Y Tam, MD, FACP, Principal Investigator — University of Toronto, Ontario, Canada
Locations (1):
- University of Toronto, Toronto, Ontario, Canada